CLINICAL TRIAL: NCT07227103
Title: A Randomized, Double-Blind Controlled Comparison of NRX-101 vs. Placebo for Adults Being Treated With Transcranial Magnetic Stimulation for Treatment Resistant Depression
Acronym: DCS_TMS
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NeuroRx, Inc. (Industry)
Collaborators: AMPA Health, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX-101_004
Expanded Access: Available
Record Dates: First submitted 2025-11-09; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matched drug and placebo capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Transcranial Magnetic Stimulation plus NRX-101 (Experimental): Participants are treated with ONE-D TMS plus NRX-101 175mg DCS/8.5mg Lurasidone once daily for five days
  Interventions: Device: ONE-D TMS; Drug: NRX-101
- Transcranial Magnetic Stimualtion (Placebo Comparator): Participants are treated with ONE-D TMS plus placebo once daily for five days
  Interventions: Device: ONE-D TMS

INTERVENTIONS:
Device: ONE-D TMS — One Day TMS Protocol performed with the AMPA TMS Device 30 Theta burst pulses delivered as per protocol
  Other Names: One Day TMS Protocol performed with the AMPA TMS Device
Drug: NRX-101 — D-cycloserine 175mg + Lurasidone 8.5mg
  Arms: Transcranial Magnetic Stimulation plus NRX-101

SUMMARY:
Major depressive disorder (MDD) is a significant public health problem and leading cause of worldwide disability. Treatment resistance is common in MDD, however, for these individuals, targeted noninvasive brain stimulation is an alternative. Repetitive transcranial magnetic stimulation (rTMS) and more recently, theta-burst stimulation (TBS), are the noninvasive brain stimulation modalities with the largest evidence base in MDD. Although efficacious, an unacceptable proportion of patients do not significantly improve, and several aspects of the TMS parameter space are under investigation to enhance clinical outcomes.

DCS has been shown in a randomized trial of more than double the percent response and remission from traditional TMS. When the AMPA one day (ONE-D) TMS protocol was combined with DCS, the measured response rate was 87% at one week.

This trial will compare response and remission at six weeks following Transcranial Magnetic Stimulation + D-cycloserine vs. TMS+placebo.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a significant public health problem and leading cause of worldwide disability. Treatment resistance is common in MDD, however, for these individuals, targeted noninvasive brain stimulation is an alternative. Repetitive transcranial magnetic stimulation (rTMS) and more recently, theta-burst stimulation (TBS), are the noninvasive brain stimulation modalities with the largest evidence base in MDD. Although efficacious, an unacceptable proportion of patients do not significantly improve, and several aspects of the TMS parameter space are under investigation to enhance clinical outcomes.

rTMS and TBS are believed to depend on synaptic plasticity in targeted circuits. Yet, there are several lines of evidence to suggest that synaptic plasticity is not intact in MDD, such as impaired learning and memory and lower expression of trophic factors.Using TMS as a tool to probe synaptic plasticity, individuals with MDD have reduced long-term potentiation-like facilitation in the motor cortex and prefrontal cortex. Importantly, this is observed with the intermittent TBS (iTBS) protocol used in MDD treatment. As such, iTBS treatment effects may be constrained by impaired synaptic plasticity in MDD.

One potential strategy to improve outcomes is to adjunctively target the N-methyl-D-aspartate (NMDA) receptor during stimulation, an ionotropic glutamate receptor and key regulator of synaptic plasticity.Synaptic plasticity with continuous and intermittent TBS is NMDA-receptor dependent, as antagonists abolish the effects of both protocols.We have shown that targeting the NMDA receptor with low doses of the partial agonist, D-cycloserine (DCS), normalizes long-term motor cortex plasticity in individuals with MDD. Moreover, it results in greater persistence of iTBS-induced changes compared with placebo.However, a demonstration that these physiological effects have an impact on treatment outcomes is needed

DCS has been shown in a randomized trial of more than double the percent response and remission from traditional TMS. When the AMPA one day (ONE-D) TMS protocol was combined with DCS, the measured response rate was 87% at one week.

This trial will compare response and remission at six weeks following Transcranial Magnetic Stimulation + D-cycloserine vs. TMS+placebo.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: A patient is eligible for inclusion in this study only if all of the following criteria apply:

  1. 18 to 65 years of age, inclusive, at Screening.
  2. Scheduled for Transcranial Magnetic Stimulation by a treating physician.
  3. Able to understand and provide written and dated informed consent prior to Screening.
  4. Deemed likely to comply with the study protocol, including communication of adverse events (AEs) and other clinically important information, including adherence to the text messaging component of the trial.
  5. Will follow medical directions for psychiatric care, as appropriate, per the standard of care.
  6. Resides in a stable living situation. A stable living situation will be defined as a minimum of 3 months at the same address with a reasonable expectation that the situation will continue such that the patient's ability to participate in the study will not be affected. Please note that housing in a shelter of any kind will not be deemed stable housing.
  7. Previously diagnosed with treatment-resistant depression according to the criteria defined in the DSM-V and having failed treatment with at least two Selective Serotonin Reuptake Inhibitor (SSRI) drugs.
  8. Has an identified reliable informant/care partner that is willing to provide information and/or supportive care as necessary.
  9. No active suicidality (without the intention to act) as evidenced by a score of 3 or less on the Columbia Suicide Severity Rating Scale.
  10. A total score greater than or equal to 25 on the 10 items of the MADRS.
  11. No co-morbidities as ascertained by medical history, physical examination (including measurement of vital signs), clinical laboratory evaluations, and electrocardiogram (ECG) which might interfere with compliance or the ability to assess efficacy or safety.
  12. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following criteria, and agrees to continue use of the same method of birth control for the duration of study participation:

      a. Non-childbearing potential: physiologically incapable of becoming pregnant (i.e., permanently sterilized [status post-hysterectomy, bilateral tubal ligation], or post-menopausal with last menses at least one year prior to Screening); or b. Childbearing potential, and meets the following criteria: i. Use of any form of hormonal birth control for at least 2 months prior to Screening, on hormone replacement therapy that started prior to 12 months of amenorrhea, using an intrauterine device (IUD) for at least 1 month prior to Screening, in a monogamous relationship with a partner who has had a vasectomy, or sexually abstinent.

      ii. Negative urinary pregnancy test at Screening, confirmed by a second negative urinary pregnancy test at Day 1, prior to receiving study treatment.
  13. Body mass index (BMI) between 18-40 kg/m2; BMI up to 45 kg/m2 is allowed with Medical Monitor review and approval.
  14. If receiving concurrent psychotherapy, the type and frequency of the therapy (e.g., weekly or monthly) has been stable for at least 3 months prior to Screening and is expected to remain stable for the duration of study participation.
  15. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, maximum 2 mg daily, or trazodone) will be allowed if the therapy has been stable for at least 4-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study.
  16. Concurrent treatment with benzodiazepines is allowed up to a maximum dose 2mg/daily used for anxiety if therapy has been stable relative to dose and schedule for at least four-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study.
  17. If women are receiving hormone replacement therapy or estrogen replacement, the therapy has been stable for at least 3 months prior to screening and is expected to remain stable for the duration of the study participation.

      Exclusion Criteria:

      Exclusion criteria: A patient is ineligible for inclusion in this study if any of the following criteria apply:

  <!-- -->

  1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
  2. Female who is pregnant or breastfeeding.
  3. Female with a positive pregnancy test at Screening or prior to randomization.
  4. Current DSM-5 diagnosis of moderate or severe substance use disorder (except marijuana or tobacco use disorder) within the 12 months prior to Screening. (Note: Substance use disorder cannot be the precipitant for study entry).
  5. A lifetime history of

     1. phencyclidine (PCP)/ketamine drug abuse, or
     2. failed use of ketamine for depression or suicidality.
  6. History of schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.
  7. History of anorexia nervosa, bulimia nervosa, eating disorder not otherwise specified (NOS), or other specified feeding and eating disorders (OSFED) within 3 years of Screening.
  8. Has dementia, delirium, amnestic, or any other cognitive disorder.
  9. Current major psychiatric disorder, diagnosed at Screening with the MINI 7.0.2 which is the primary focus of treatment, with bipolar disorder as the secondary focus of treatment, within the past 6 months.
  10. Estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m2 using the Cockcroft-Gault formula.
  11. A clinically significant abnormality on the Screening physical examination that may affect safety or study participation, or that may confound interpretation of study results according to the study clinician.
  12. Current episode of:

      1. Myocardial infarction within 1 year of Screening.
      2. Diagnosis of angina pectoris.
      3. Prolonged QTc interval, as measured by Fridericia's correction formula (QTcF) ≥450 msec at Screening for males or ≥ 470 msec for females on 2 of 3 measurements at least 15 minutes apart prior to randomization on Day 1.
  13. Diagnosis of chronic lung disease, excluding asthma.
  14. Lifetime history of any of the following: surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's Disease, Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the clinician, is deemed associated with significant injury to, or malfunction of, the CNS.
  15. History of significant head trauma within the past two years.
  16. Diabetes mellitus fulfilling any of the following criteria:

      1. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.0 percent at Screening.
      2. Admitted to the hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.
      3. Not under physician care for diabetes mellitus.
      4. Not on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to Screening.
      5. Not on the same dose of oral thiazolidinediones (glitazones) for the 8 weeks prior to Screening.
  17. Any current or past history of any physical condition which, in the opinion of the investigator, may put the patient at risk or interfere with study results interpretation.
  18. Diagnosis of HIV/AIDS.
  19. Diagnosis of Hepatitis C.
  20. On exclusionary concomitant psychotropic and non-psychotropic medications (see Appendix 1).
  21. Prescribed more than one agent in each of the following categories at randomization:

      1. Approved SSRIs.
      2. Approved serotonin and norepinephrine reuptake inhibitors (SNRIs).
      3. Approved tetracyclic antidepressants (TeCAs).
  22. Currently prescribed oxcarbazepine or carbamazepine.
  23. Exclusionary laboratory values or any other clinically significant abnormal laboratory result at Screening. Within normal limits (WNL) will be determined based on lab values of the local lab used.
  24. Known allergies to lurasidone or Latuda®, cycloserine or Seromycin®, or the following excipients: mannitol, croscarmellose sodium, magnesium stearate, silicon dioxide, and/or hydroxypropylmethylcellulose (HPMC).
  25. Participation in any clinical trial with an investigational drug or device within the past month or planned concurrent study participation.
  26. Study site personnel and/or persons employed by NRx Pharma, Inc., the Contract Research Organization (CRO), the investigator, or study site (i.e., permanent, temporary contract worker, or designee responsible for the conduct of the study), or an immediate family member (i.e., spouse, parent, child, or sibling [biological or legally adopted]) of such persons.
  27. Positive urine toxicity screening for use of any cocaine, opiates, non-prescribed amphetamines, or non-prescribed barbiturates. (Note: cannabinoids or marijuana use is not exclusionary, unless patient meets the DSM-5 criteria for cannabis withdrawal).
  28. Signs and symptoms of active or residual COVID-19, or unresolved symptoms of COVID-19 that impact health, e.g. requirements for oxygen supplementation, etc. Discharged from an inpatient hospitalization for more than 48 hours for COVID-19 within the past 28 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
MADRS Depression | 6 weeks
  Montgomery Asberg Depression Rating Scale Total Score
CGI-SS Suicidality | 6 weeks
  Clinical Global Impression Suicidality Scale

SECONDARY OUTCOMES:
Percent Response | Six weeks
  Percent Response from Depression
Percent Remission from Depression | Six weeks
  Percent Remission from Depression
Percent Remission from Suicidality | Six weeks
  Percent Remission from Suicidality
Percent Improvement on EMOBOT | Six weeks
  Percent improvement on EMOBOT phone app

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen and Associates, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes